CLINICAL TRIAL: NCT03821116
Title: Milk and Soured Milk (filmjölk) Intervention on Oxidative Stress and Inflammation: A Randomized Crossover Intervention Study
Brief Title: Milk and Soured Milk (filmjölk) Intervention on Oxidative Stress and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Forte (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MILK: EPN-Uppsala dnr 2018-328
Record Dates: First submitted 2019-01-16; First posted 2019-01-29 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Oxidative Stress; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milk (Experimental): At least 500 ml of Swedish milk daily for three weeks (crossover). Intervention and crossover preceded by 3 weeks with max 50 ml of milk or soured milk (filmjölk) daily. Fat content of milk and soured milk should be the same: 0.5%, 1.5% or 3%.
  Interventions: Other: Milk
- Soured milk (filmjölk) (Experimental): At least 500 ml of Swedish soured milk (filmjölk) daily for three weeks (crossover). Intervention and crossover preceded by 3 weeks with max 50 ml of milk or soured milk (filmjölk) daily. Fat content of milk and soured milk should be the same: 0.5%, 1.5% or 3%.
  Interventions: Other: Soured milk (filmjölk)

INTERVENTIONS:
Other: Milk — Swedish milk from cow.
  Arms: Milk
Other: Soured milk (filmjölk) — Swedish soured milk (from cow milk).
  Arms: Soured milk (filmjölk)

SUMMARY:
This study evaluates a high intake of milk compared with a high intake of soured milk (Swedish filmjölk) on markers of oxidative stress and inflammation in a randomized crossover intervention study.

DETAILED DESCRIPTION:
A diet rich in antioxidants reduces oxidative stress and inflammation and could potentially improve health and lower the rate of hip fracture. Milk and dairy are also promoted as part of a healthy diet since they contain 18 of 22 essential nutrients including calcium, phosphorous, and vitamin D and have been suggested to be associated with lower risk of cardiovascular disease, especially stroke, type 2 diabetes, and cancer. Meta-analyses of milk and dairy on fracture and mortality risk in cohort studies are, however, inconclusive and show significant heterogeneity between studies. Small intakes may have beneficial effects in comparison to null intake whereas higher intakes may have other effects and non-linear relationships are rarely examined. Frequently, different milk products are considered as one entity in cohort studies. The investigators recently showed that different milk products might have differential effects on disease. A high long-term milk intake was associated with an increased risk of mortality (total, cardiovascular, and cancer mortality) and hip fracture, especially among women, whereas a high long-term intake of fermented milk (soured milk and yogurt or cheese) was associated with a lower risk of mortality and fracture among women. Similar results have been presented for total mortality (Northern Sweden) and humeral fractures (South-Eastern Australia).

Intake of milk and fermented milk is of tradition high in Sweden. The prevalence of lactase persistence is high (around 95%). The range in milk intake from non- and low-consumers to high consumers makes Sweden an appropriate setting for epidemiological and interventional studies.

A common potential mechanism for intake of fruits, vegetables, and different dairy products on risk of disease is their influence on inflammation and oxidative stress. Chronic low-grade inflammation and age-related increase of oxidative stress are suggested pathogenic mechanisms of premature ageing and many diseases including cardiovascular disease, cancer, accelerated bone loss (leading to osteoporosis), and age-related reduction of muscle strength and mass (sarcopenia) with potential impacts on risk of falling and fracture. The lower risk of fractures with a high intake of fermented milk products observed may be due to potential probiotic, antioxidative, and anti-inflammatory effects and effects on gut microbiota. A high intake of milk was not only associated with risk of mortality and fractures but also with increased concentrations of inflammation and oxidative stress markers. An inverse association was seen for intake of soured milk and yogurt [Michaëlsson, 2014]. Fermented milk products with probiotics have been shown to reduce the levels of inflammation markers, other studies have been small to show conclusive effects and results may also be dependent on the probiotic strain. A head-to-head comparison of the effect of regular milk and soured milk (or yogurt) on markers of inflammation and oxidative stress in a randomized intervention study is warranted. The randomized crossover intervention study will be performed among both men and women.

The aim of the study is to examine the potentially different short-term effects of milk and sour milk on markers of oxidative stress and inflammation in a randomized cross-over trial. The research questions are:

1. In a randomized cross-over trial, what is the effect of a daily intake of at least 500 ml of Swedish milk compared with an intake of at least 500 ml Swedish soured milk (filmjölk) during 3 weeks on markers of oxidative stress and inflammation?
2. What are the effects of these milk products on a large number of proteins related with inflammation and ageing diseases, assessed with large-scale proteomic analysis?
3. What are the effects of these milk products on metabolites involved in inflammation and ageing diseases using large-scale metabolomics analysis?
4. What are the effects of these milk products on the gut microflora (microbiome)?

Changes in proteomics, metabolomics and the gut microbiome are other pre-specified outcome measures but since they are exploratory in nature, we do not specify them under outcomes since it is not possible to exactly specify these outcome measures. Exploratory analyses will include whether effects are different between men and women, dependent on body composition (assessed with whole body dual X-ray absorptiometry, DXA) or long-term dietary intake (assessed by fatty acid composition in subcutaneous fat). Participants will be allowed to consume more than 500 ml of milk/filmjölk during the intervention periods and, if possible, a potential dose-response effect will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Tolerates both a low and a high intake of milk and soured milk
* Agrees to comply with study protocol

Exclusion Criteria:

* Inflammatory bowel disease
* Major gastric tract operation
* Pregnancy
* Eating disorder

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Change in oxidative stress marker | baseline and 3 weeks
  urinary 8-iso-prostaglandin F2 alpha (8-iso-PGF2alpha)
Change in oxidative stress marker | 6 weeks and 9 weeks
  urinary 8-iso-prostaglandin F2 alpha (8-iso-PGF2alpha)

SECONDARY OUTCOMES:
Change in interleukin-6 (IL-6) | baseline and 3 weeks
  Inflammation marker, measured in serum
Change in interleukin-6 (IL-6) | 6 weeks and 9 weeks
  Inflammation marker, measured in serum
Change high sensitive C-reactive protein (hs-CRP) | baseline and 3 weeks
  Inflammation marker, measured in serum
Change high sensitive C-reactive protein (hs-CRP) | 6 weeks and 9 weeks
  Inflammation marker, measured in serum
Change in 15-keto-dihydro-prostaglandin F2 alpha (15-keto-dihydro-PGF2alpha) | baseline and 3 weeks
  Inflammation marker, a major metabolite of prostaglandin F2alpha, measured in urine
Change in 15-keto-dihydro-prostaglandin F2 alpha (15-keto-dihydro-PGF2alpha) | 6 weeks and 9 weeks
  Inflammation marker, a major metabolite of prostaglandin F2alpha, measured in urine

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Byberg, PhD, Principal Investigator — Department of Surgical Sciences, Uppsala University
Locations (1):
- Forskningsmottagning bentäthet, Kirurgiska vetenskaper, Uppsala Universitet, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larsson SC, Crippa A, Orsini N, Wolk A, Michaelsson K. Milk Consumption and Mortality from All Causes, Cardiovascular Disease, and Cancer: A Systematic Review and Meta-Analysis. Nutrients. 2015 Sep 11;7(9):7749-63. doi: 10.3390/nu7095363. PMID 26378576
- [Background] Michaelsson K, Wolk A, Langenskiold S, Basu S, Warensjo Lemming E, Melhus H, Byberg L. Milk intake and risk of mortality and fractures in women and men: cohort studies. BMJ. 2014 Oct 28;349:g6015. doi: 10.1136/bmj.g6015. PMID 25352269
- [Background] Tognon G, Nilsson LM, Shungin D, Lissner L, Jansson JH, Renstrom F, Wennberg M, Winkvist A, Johansson I. Nonfermented milk and other dairy products: associations with all-cause mortality. Am J Clin Nutr. 2017 Jun;105(6):1502-1511. doi: 10.3945/ajcn.116.140798. Epub 2017 May 10. PMID 28490510
- [Background] Holloway KL, Bucki-Smith G, Morse AG, Brennan-Olsen SL, Kotowicz MA, Moloney DJ, Sanders KM, Korn S, Timney EN, Dobbins AG, Pasco JA. Humeral Fractures in South-Eastern Australia: Epidemiology and Risk Factors. Calcif Tissue Int. 2015 Nov;97(5):453-65. doi: 10.1007/s00223-015-0039-9. Epub 2015 Jul 14. PMID 26169198